CLINICAL TRIAL: NCT04891250
Title: The Zambia Ivermectin Trial for the Treatment and Prevention of COVID-19
Acronym: ZIT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Collaborators: Ministry of Health, Zambia (Other Government); University of Zambia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZIT
Record Dates: First submitted 2021-05-11; First posted 2021-05-18 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: SARS-CoV-2; Ivermectin
MeSH Terms: interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: Patients with moderate to severe COVID-19 disease will be randomized to either Ivermectin (Intervention) or Standard of Care (Control arm) in a 1:1 ratio.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Patients with moderate to severe COVID-19 disease will be randomized to either Ivermectin (Intervention) or Standard of Care (Control arm) in a 1:1 ratio
  Interventions: Drug: Ivermectin
- Prophylaxis (Experimental): An additional group of patients will be recruited will be randomized to either Ivermectin as prophylaxis (Intervention) or Standard of Care with no ivermectin (Control arm) in a 1:1 ratio
  Interventions: Other: Prophylaxis

INTERVENTIONS:
Drug: Ivermectin — Treatment of SARS Cov-2 patients with Ivermectin
  Arms: Intervention
Other: Prophylaxis — Treatment of high risk population with Ivermectin as prophylaxis
  Arms: Prophylaxis

SUMMARY:
The study aims to test whether Ivermectin would decrease mortality and reduces chances of getting infected with corona virus, improve management of clinical symptoms and reduce length of stay in ICU and transition probabilities to ICU (ventilator).

DETAILED DESCRIPTION:
With the onset of global pandemic of the Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) and the sharp rise in infection and mortality rates, efficient management of the current medical emergency has become an absolute priority. A lot of resources have been directed to developing a comprehensive therapeutic approach to preventing and curing this disease, and this has mostly been in western countries. However, lack of definite treatment, high number of infected people, limited capacity and the impact of COVID-19 on existing health infrastructure has left biomedical researchers and clinicians faced with the mammoth task of providing appropriate clinical care solutions and strategies with favorable cost-benefit outcomes, which can help in both curbing the disease and treating patients. To meet this challenge, repurposing of available drugs has become vital. Evidence from several recent clinical trials on the effects of available therapeutic clinical drugs and vitamin supplements on mortality rate and other clinical outcomes associated with COVID-19 are promising, however, the efficacy, safety, and appropriate dosing of therapeutic clinical drugs such as ivermectin, remain largely unevaluated in Sub-Saharan Africa. The investigators propose to evaluate and compare the efficacy of ivermectin in the management of Covid-19.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed positive for SARS-CoV-2 by real-time reverse transcription PCR (rRT-PCR with presence of a fever, cough, and/or sore throat.

Exclusion Criteria:

* Patients will be excluded if they report to be allergic to ivermectin or if there is potential for a drug-drug interaction with ivermectin;
* Have chronic illnesses (e.g., ischemic heart disease, heart failure, documented cardiomyopathy, chronic kidney disease, chronic liver disease);
* Have received ivermectin in the last 7 days; are pregnant or lactating;
* Or have participated in any other clinical trial within the last month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
All-cause COVID-19 related mortality | within 28 days of enrollment
  All-cause COVID-19 related mortality
COVID-19 Infection | Study duration
  the proportion of patients on Ivermectin prophylaxis who test positive for COVID 19 using PCR after initially testing negative at enrolment

SECONDARY OUTCOMES:
Patient cure rate | 14- 28 days
  The percentage of cured patients, defined as symptoms free to be discharged from the hospital and the percentage Changes of WHO's OSCI scale for COVID-19 between baseline and day 14 and between baseline and day 28. The study will will also evaluate the time to cure in both groups by measuring time from admission of the patient to the hospital till discharge.
Participant Infection Rate | 90 days
  determine proportion who will develop severe disease and needing admission in addition to the above outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zambia, Lusaka, Zambia

REFERENCES:
- [Background] Annweiler C, Beaudenon M, Gautier J, Simon R, Dubee V, Gonsard J, Parot-Schinkel E; COVIT-TRIAL study group. COvid-19 and high-dose VITamin D supplementation TRIAL in high-risk older patients (COVIT-TRIAL): study protocol for a randomized controlled trial. Trials. 2020 Dec 28;21(1):1031. doi: 10.1186/s13063-020-04928-5. PMID 33371905
- [Background] Jovanovic A, Klimek P, Renn O, Schneider R, Oien K, Brown J, DiGennaro M, Liu Y, Pfau V, Jelic M, Rosen T, Caillard B, Chakravarty S, Chhantyal P. Assessing resilience of healthcare infrastructure exposed to COVID-19: emerging risks, resilience indicators, interdependencies and international standards. Environ Syst Decis. 2020;40(2):252-286. doi: 10.1007/s10669-020-09779-8. Epub 2020 Jun 4. PMID 32837821
- [Background] Chaccour C, Casellas A, Blanco-Di Matteo A, Pineda I, Fernandez-Montero A, Ruiz-Castillo P, Richardson MA, Rodriguez-Mateos M, Jordan-Iborra C, Brew J, Carmona-Torre F, Giraldez M, Laso E, Gabaldon-Figueira JC, Dobano C, Moncunill G, Yuste JR, Del Pozo JL, Rabinovich NR, Schoning V, Hammann F, Reina G, Sadaba B, Fernandez-Alonso M. The effect of early treatment with ivermectin on viral load, symptoms and humoral response in patients with non-severe COVID-19: A pilot, double-blind, placebo-controlled, randomized clinical trial. EClinicalMedicine. 2021 Feb;32:100720. doi: 10.1016/j.eclinm.2020.100720. Epub 2021 Jan 19. PMID 33495752
- [Background] Caly L, Druce JD, Catton MG, Jans DA, Wagstaff KM. The FDA-approved drug ivermectin inhibits the replication of SARS-CoV-2 in vitro. Antiviral Res. 2020 Jun;178:104787. doi: 10.1016/j.antiviral.2020.104787. Epub 2020 Apr 3. PMID 32251768
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Sevestre J, Mailhe M, Doudier B, Aubry C, Amrane S, Seng P, Hocquart M, Eldin C, Finance J, Vieira VE, Tissot-Dupont HT, Honore S, Stein A, Million M, Colson P, La Scola B, Veit V, Jacquier A, Deharo JC, Drancourt M, Fournier PE, Rolain JM, Brouqui P, Raoult D. Clinical and microbiological effect of a combination of hydroxychloroquine and azithromycin in 80 COVID-19 patients with at least a six-day follow up: A pilot observational study. Travel Med Infect Dis. 2020 Mar-Apr;34:101663. doi: 10.1016/j.tmaid.2020.101663. Epub 2020 Apr 11. PMID 32289548
- [Background] Heidary F, Gharebaghi R. Ivermectin: a systematic review from antiviral effects to COVID-19 complementary regimen. J Antibiot (Tokyo). 2020 Sep;73(9):593-602. doi: 10.1038/s41429-020-0336-z. Epub 2020 Jun 12. PMID 32533071
- [Background] Ahmed S, Karim MM, Ross AG, Hossain MS, Clemens JD, Sumiya MK, Phru CS, Rahman M, Zaman K, Somani J, Yasmin R, Hasnat MA, Kabir A, Aziz AB, Khan WA. A five-day course of ivermectin for the treatment of COVID-19 may reduce the duration of illness. Int J Infect Dis. 2021 Feb;103:214-216. doi: 10.1016/j.ijid.2020.11.191. Epub 2020 Dec 2. PMID 33278625
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204